CLINICAL TRIAL: NCT05197933
Title: Safety of Laparoscopic Resection for Gastrointestinal Stromal Tumor on Unfavorable Anatomic Site of Stomach：a Multicenter Prospective Trial（CLASS-06）
Brief Title: Safety of Laparoscopic Resection for Gastrointestinal Stromal Tumor on Unfavorable Anatomic Site of Stomach
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other); Peking University Cancer Hospital & Institute (Other); Shanghai Zhongshan Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Fujian Medical University Union Hospital (Other); Peking University People's Hospital (Other); Ruijin Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); West China Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Liaoning Cancer Hospital & Institute (Other); Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Hui Cao, Professor, RenJi Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLASS-06
Record Dates: First submitted 2021-09-07; First posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: Gastrointestinal Stromal Tumors; Unfavorable Anatomic Site of Stomach; Laparoscopic Resection
MeSH Terms: conditions — Gastrointestinal Stromal Tumors

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, open-label, single-arm
Masking Description: Blinding Method: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laparoscopic resection (Experimental): laparoscopic resection for GIST at unfavorable anatomic sites of stomach
  Interventions: Procedure: Laparoscopic resection

INTERVENTIONS:
Procedure: Laparoscopic resection — Laparoscopic resection for GIST at unfavorable anatomic site of stomach will be conducted

SUMMARY:
The aim of this trial is to evaluate the safety of laparoscopic resection for GIST whose diameter is ≥2cm and ≤5cm at unfavorable anatomic sites of stomach.

DETAILED DESCRIPTION:
The aim of this trial is to evaluate the safety of laparoscopic resection for GIST whose diameter is ≥2cm and ≤5cm at unfavorable anatomic sites of stomach. Unfavorable anatomic sites are defined by soft tissue sarcoma, NCCN Clinical Practice Guidelines in Oncology (version 2. 2018). The defined laparoscopy unfavorable sites including the anatomic sites of stomach other than greater curvature and front wall, including the less curvature, the posterior wall, and adjacent to cardia and pylorus.

ELIGIBILITY:
Inclusion Criteria:

* Age from over 18 to under 75 years;
* Gastrointestinal stromal tumor at unfavorable anatomic sites of stomach preoperatively confirmed by endoscopy, ultrasound endoscopy, CT or MRI;
* Diameter of tumor size is ≥2cm and ≤5cm confirmed by contrast CT or MRI;
* Patients whose tumor is resectable by laparoscopic technique at preoperative assessment;
* No evidence of distant metastasis and tumor invading nearby organs at preoperative assessment;
* Performance status of 0 or 1 on ECOG (Eastern Cooperative Oncology Group) scale;
* ASA (American Society of Anesthesiology) score I, II, or III;
* Written informed consent.

Exclusion Criteria:

* Women during pregnancy or breast-feeding;
* Severe mental disorder;
* History of previous upper abdominal surgery (except laparoscopic cholecystectomy);
* History of other malignant disease within the past five years;
* History of previous neoadjuvant imatinib therapy;
* History of unstable angina or myocardial infarction within the past six months;
* History of cerebrovascular accident within the past six months;
* History of continuous systematic administration of corticosteroids within the past month;
* Requirement of simultaneous surgery for other disease;
* Emergency surgery due to complication (bleeding, obstruction or perforation) caused by gastrointestinal stromal tumor;
* FEV1<50% of predicted value;
* Patients with GIST locates at favorable anatomic sites detected by contrast CT, MRI or ultrasound endoscopy at preoperative assessment;
* Patients with GIST diameter<2cm or>5cm detected by contrast CT or MRI;
* Presence of distant metastasis or tumor invading nearby organs at preoperative assessment.

Withdrawal Criteria:

* Patients postoperatively confirmed as non-GIST case by pathology (These cases are enrolled in safe group for future statistic analysis);
* GIST at unfavorable anatomic site diagnosed before operation, while GIST at favorable anatomic site determined by intraoperative exploration;
* Patients confirmed as tumor rupture , metastasis or invading nearby organs intraoperately;
* Patients requiring simultaneous surgical treatment of other diseases;
* Sudden severe complications during the perioperative period (intolerable surgery or anesthesia), which renders it unsuitable or unfeasible to implement the study treatment protocol as scheduled;
* Patients confirmed to require emergency surgery by attending physicians due to changes in the patient's condition after inclusion in this study;
* Patients who voluntarily quit or discontinue treatment for personal reasons at any stage after inclusion in this study;
* Treatment implemented is proven to violate study protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
3-year disease-free survival rate (DFS) | until the date of first documented progression, assessed up to 3 years
  The number of patients with DFS > 3 years was used as the numerator and the number of all patients was used as the denominator to calculate the ratio value.

SECONDARY OUTCOMES:
Success rate of laparoscopic surgery | postoperative 15 days
  The proportion value will be calculated for the number of patients receiving laparoscopic local resection for GIST locating at unfavorable sites of stomach and meet the following 4 criteria as the numerator and the number of all patient undergo surgical treatment (laparoscopic surgery/laparotomy) as the denominator.
  Definition of successful laparoscopic resection：
  。① Resection is completed by total laparoscopy (extra auxiliary incision is not required. Tumor is extracted through the extended trocar incision)；②Tumor is completely resected without rupture which complys with the principle of tumor isolation；③No conversion from laparoscopy to laparotomy due to incidences that laparascopy can not complete, including hemorrhage, unresectable tumor etc；④Resected margin confirmed to be negative by postoperative pathology.
  All the previous 4 criteria have to be achieved simultaneously to be considered a complete laparoscopic surgery.
Rate of intraoperative complication | intraoperative time
  The proportion value will be calculated for the number of patients with any intraoperative complication as the numerator and the number of all patients undergoing surgical treatment (laparoscopic surgery/laparotomy) as the denominator.
Rate of Postoperative complication | postoperative 30 days, or the discharge day if hospitalization>30 days
  The proportion value will be calculated for the number of patients with any postoperative complication as the numerator and the number of all patients undergoing surgical treatment (laparoscopic surgery/laparotomy) as the denominator.
3-year overall survival rate (OS) | until the date of first documented progression, assessed up to 3 years
  The number of patients with OS > 3 years was used as the numerator and the number of all patients was used as the denominator to calculate the ratio value.
Postoperative recovery course（Time to start off-bed activities, bowel function, to restore liquid food and semi-liquid food） | postoperative 30 days, or the discharge day if hospitalization>30 days
  Time to start off-bed activities, bowel function, to restore liquid food and semi-liquid food
  * Starting from the postoperative day 1 to the first postoperative discharge, within the initial recognition of the earliest time for off-bed activities, bowel function (flatulence/bowel movement), to restoration of fluid/semi-fluid diet; records are made hourly.
  * Flatulence/bowel movement on the day of surgery is excluded.
  * In case of no off-bed activities/flatulence/bowel movement/restoration of liquid/semi-liquid diet before the first postoperative discharge, the discharge time should be recorded as the time of off-bed activities/flatulence/bowel movement/restoration of liquid/semi-liquid diet.
  * The initial time of off-bed activities/flatulence/bowel movement/restoration of liquid/semi-liquid diet is per patient report.
Postoperative recovery course（Highest Body Temperature） | postoperative 3 days
  Highest Body Temperature
  • The highest body temperature starting from postoperative day 1 up to day 3 should be measured at least three times a day.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Cao, Professor, Study Chair — RenJi Hospital
Locations (1):
- Renji hospital, Shanghai, Shanghai Municipality, China

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT05197933/Prot_SAP_ICF_000.pdf